CLINICAL TRIAL: NCT03324321
Title: Feasibility of Improving Cerebral Autoregulation in Acute Intracerebral Haemorrhage (BREATHE-ICH) Study
Brief Title: Feasibility of Improving Cerebral Autoregulation in Acute Intracerebral Haemorrhage
Acronym: BREATHE-ICH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Leicester (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 0624
Record Dates: First submitted 2017-10-09; First posted 2017-10-27 (Actual); Last update posted 2018-10-31 (Actual); Status verified 2018-10

CONDITIONS: Stroke, Acute; Hemorrhage; Cerebral Brain Hemorrhage; Blood Pressure
Keywords: Cerebral Haemodynamics; Carbon Dioxide; Cerebral Autoregulation
MeSH Terms: conditions — Stroke; Hemorrhage; Cerebral Hemorrhage

STUDY DESIGN:
Intervention Model Description: Single-centre, prospective, before and after study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hyperventilation Protocol (Experimental): This will involve sustained periods of 90-seconds of hyperventilation at two levels (-5mmHg and -10mmHg below baseline EtCO2) to a maximum lower level threshold of EtCO2 24mmHg/CBFV 33cm/s regulated using a metronome. Two-minute washout periods of normal respiration will be allowed between successive measurements. Each incremental reduction in pCO2 will be repeated on two occasions during the same session. Further assessments will be conducted 10-14 days following baseline assessments.
  Interventions: Other: Hypocapnia via Hyperventilation Protocol

INTERVENTIONS:
Other: Hypocapnia via Hyperventilation Protocol — 90 seconds of hyperventilation using a metronome to lower levels of -5mmHg and -10mmHg below baseline EtCO2

SUMMARY:
In the UK, 23,000 (15%) of the 150,000 people who suffer a stroke each year have bleeding in the brain, also referred to as acute intracerebral haemorrhage (ICH). An Autoregulation Index (ARI) can be assigned between 0 and 9 (0 being poor and 9 being the most efficient CA observed) to gauge how good the control over blood flow is at a given time. Dynamic CA (dCA) is a measure of the response of cerebral blood flow (CBF) to rapid changes in blood pressure (BP), and several key studies have shown impaired dCA post-acute ICH. The most recent study demonstrated that dCA impairment lasts up to 12 days. This is particularly important to understand, since our preliminary work has recently shown that changes in carbon dioxide using simple breathing exercises can improve Autoregulation.

Unfortunately, there are limited non-pharmacological management options and significant opportunities to improve patient outcome in ICH. The proposed study addresses this area, by investigating whether a simple breathing exercise in survivors of ICH is safe, feasible and effective in reducing brain injury by improving cerebral autoregulation.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of a haemorrhagic stroke within 48 hours of onset (for patients waking with a stroke, time of onset will be taken to be the time when the patient was last asymptomatic)
* Able and willing to give informed consent
* Male or female, aged 18 years or above
* Able (in the Investigator's opinion) and willing to comply with all study requirements
* Willing to allow his or her General Practitioner (GP) to be notified of participation in the study

Exclusion Criteria:

* Male or Female, aged under 18 years
* Significant previous airways disease (formal diagnosis of moderate or severe airways disease and having treatment for this respiratory condition - via inhalers or specialist input)
* Unable (in the Investigator's opinion) or unwilling to comply with any study requirements
* Female participants who are pregnant, lactating or planning pregnancy during the course of the study
* Clinical diagnosis of stroke greater than 48 hours from onset
* Having had a resolved transient ischaemic attack (TIA) (i.e. neurological symptoms completely resolved upon hospital presentation)
* Co-morbidity with anticipated life expectancy less than 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2017-10-08 (Actual); Primary Completion 2018-07-15 (Actual); Study Completion 2018-07-15 (Actual)

PRIMARY OUTCOMES:
Post Stroke Morbidity and Mortality | 14 days
  Determined using Modified Rankin Scale 0 - No symptoms
  1. - No significant disability, despite symptoms; able to perform all usual duties and activities
  2. - Slight disability; unable to perform all previous activities but able to look after own affairs without assistance
  3. - Moderate disability; requires some help, but able to walk without assistance
  4. - Moderate severe disability; unable to walk without assistance and unable to attend to own bodily needs without assistance
  5. - Severe disability; bedridden, incontinent, and requires constant care 6- Death
The percentage of recruited subjects able to comply with the full measurement protocol | 14 days
The percentage of measurements rejected because of aspects related to data quality during the analysis protocol, with recorded reasons | 14 days
The percentage of recruited subjects in whom values for the following cerebral haemodynamic parameters can be derived | 14 days
  * % change in CBFv at baseline and in response to a hyperventilation manoeuvre in the acute (<48 hours) and sub-acute (10 to 14 days) periods
  * Autoregulation index
    * % change in CBFv at baseline and in response to a hyperventilation manoeuvre in the acute (<48 hours) and sub-acute (10 to 14 days) periods
    * Autoregulation index

CONTACTS AND LOCATIONS:
Overall Officials: Thompson G Robinson, MD, FRCP, Principal Investigator — University of Leicester
Locations (1):
- University Hospitals of Leicester NHS Trust, Leicester, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tiecks FP, Lam AM, Aaslid R, Newell DW. Comparison of static and dynamic cerebral autoregulation measurements. Stroke. 1995 Jun;26(6):1014-9. doi: 10.1161/01.str.26.6.1014. PMID 7762016
- [Background] Ma H, Guo ZN, Liu J, Xing Y, Zhao R, Yang Y. Temporal Course of Dynamic Cerebral Autoregulation in Patients With Intracerebral Hemorrhage. Stroke. 2016 Mar;47(3):674-81. doi: 10.1161/STROKEAHA.115.011453. Epub 2016 Feb 4. PMID 26846864
- [Derived] Minhas JS, Panerai RB, Swienton D, Robinson TG. Feasibility of improving cerebral autoregulation in acute intracerebral hemorrhage (BREATHE-ICH) study: Results from an experimental interventional study. Int J Stroke. 2020 Aug;15(6):627-637. doi: 10.1177/1747493019873690. Epub 2019 Sep 9. PMID 31500552
- [Derived] Minhas JS, Panerai RB, Robinson TG. Feasibility of Improving Cerebral Autoregulation in Acute Intracerebral Haemorrhage (BREATHE-ICH) study: a protocol for an experimental interventional study. BMJ Open. 2018 Mar 27;8(3):e020758. doi: 10.1136/bmjopen-2017-020758. PMID 29593024
- Available data/document: Funder — http://dunhillmedical.org.uk/ — Dunhill RTF Grant (RTF97/0117)